CLINICAL TRIAL: NCT00539266
Title: Autologous Bone Marrow-derived Mononuclear Cells for Therapeutic Arteriogenesis in Patients With Limb Ischemia A Double Blind, Placebo Controlled, Study in Diabetic and Non-diabetic Patients
Brief Title: Autologous Bone Marrow-derived Mononuclear Cells for Therapeutic Arteriogenesis in Patients With Limb Ischemia
Acronym: ABC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Board of Directors, Leiden University Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P07.058
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2007-10

CONDITIONS: Intermittent Claudication; Peripheral Vascular Diseases
Keywords: Claudication; Critical limb ischemia; Cell therapy; Bone marrow
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): non diabetic patients with Fontaine IIb-IV peripheral artery disease
  Interventions: Biological: bone marrow derived mononuclear cells
- 2 (Placebo Comparator): non diabetic patients with Fontaine IIb-IV peripheral artery disease
  Interventions: Biological: placebo
- 3 (Active Comparator): diabetic patients with Fontaine IIb-IV peripheral artery disease
  Interventions: Biological: bone marrow derived mononuclear cells
- 4 (Placebo Comparator): diabetic patients with Fontaine IIb-IV peripheral artery disease
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: bone marrow derived mononuclear cells — 40 IM injections (calf muscle) of 1-8 10E9 mono nuclear cells
  Arms: 1; 3
Biological: placebo — 40 IM injections (calf muscle) of placebo suspension
  Arms: 2; 4

SUMMARY:
The investigators propose confirm and extend the findings of open studies on the apparent efficacy of bone-marrow derived mononuclear cells for the induction of arteriogenesis in patients with severe claudication or critical leg ischemia and pay special attention to the influence of diabetic disease on the outcome of the study and to the possible pro-atherogenic/ pro-inflammatory effects of BM-MNC injections.

DETAILED DESCRIPTION:
Although the safety and beneficial effects of intramuscular transplantation of bone marrow derived mononuclear cells procedure appear well documented, a number of critical question regarding application of BM-MNC for peripheral vascular disease remain to be answered. First, although the original study has been partially performed as semi-blinded study (patients with double sided claudication were recruited and blindly treated with BM-MNC in one leg and peripheral blood injections in the other leg), this approach does exclude a placebo effect. Second, although patients with mild diabetes were included in the protocol, the results for diabetic patients were not analyzed separately. Diabetic disease is characterized by monocyte and endothelial progenitor cell dysfunction and it is still unclear whether this approach is also effective in diabetic patients. Third, although six-month results are reported long-term efficacy has not been established yet.

To address these issues, the investigators now propose confirm and extend the findings from open studies in a randomized double-blind study in patients with severe claudication or critical leg ischemia and pay special attention to the influence of diabetic disease on the outcome of the study and to the possible pro-atherogenic/ pro-inflammatory effects of BM-MNC injections.

ELIGIBILITY:
Inclusion Criteria:

* persistent (>3 months) disabling claudication (Fontaine's stages IIb or Rutherford's categories 3, viz. pain free walking distance less than 100 meter) despite optimal therapy or critical limb ischemia (Fontaine's stages III/IV or Rutherford's categories 4-6)
* ineligibility for angioplasty or bypass procedures
* male of female, >18 years old
* life expectancy > 1 year
* written informed consent

Exclusion Criteria:

* candidates for angioplasty or bypass procedures
* inability to undergo bone marrow harvesting
* any condition in the affected limb that is anticipated to require surgical intervention in the first weeks after BM-MNC treatment
* life threatening co-morbidity
* poorly controlled diabetes (HbA1C > 10%)
* active malignancy in the 5 years prior to treatment
* INR >1.5 at the time of bone-marrow harvest
* bleeding diathesis
* inability to undergo arterial catheterization
* inability to follow the protocol and to comply with the follow up requirements
* any other conditions that, in the opinion of the investigators, could interfere with the therapy or could pose a significant threat to the subject if the investigational therapy was to be initiated

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2007-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Limb salvage/wound healing at t=6 months; Pain free walking distance | 6 months

SECONDARY OUTCOMES:
quality of life (RAND-36), pain Scores (Brief Pain Inventory), tcO2 (wrist/ankle ratio) ABI Collateral artery scores (angiogram) at t=6 months, Limb salvage/wound healing at t= 3 and 12 months, Pain free walking distance at t=3 and 12 months, | 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan HN Lindeman, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Moazzami B, Mohammadpour Z, Zabala ZE, Farokhi E, Roohi A, Dolmatova E, Moazzami K. Local intramuscular transplantation of autologous bone marrow mononuclear cells for critical lower limb ischaemia. Cochrane Database Syst Rev. 2022 Jul 8;7(7):CD008347. doi: 10.1002/14651858.CD008347.pub4. PMID 35802393
- [Derived] Lindeman JHN, Zwaginga JJ, Kallenberg-Lantrua G, van Wissen RC, Schepers A, van Bockel HJ, Fibbe WE, Hamming JF. No Clinical Benefit of Intramuscular Delivery of Bone Marrow-derived Mononuclear Cells in Nonreconstructable Peripheral Arterial Disease: Results of a Phase-III Randomized-controlled Trial. Ann Surg. 2018 Nov;268(5):756-761. doi: 10.1097/SLA.0000000000002896. PMID 30004916